CLINICAL TRIAL: NCT06455683
Title: The Effect of Glaucoma Surgery on Aqueous Dynamics in Patients With Glaucoma or Ocular Hypertension
Brief Title: The A D A G I O Study
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 333763
Record Dates: First submitted 2024-05-28; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glaucoma: Glaucoma or Ocular Hypertension patients with sub-optimal intraocular pressure (IOP) on multiple topical medications
  Interventions: Procedure: Glaucoma Surgery

INTERVENTIONS:
Procedure: Glaucoma Surgery — One of 5 Types of Interventions will be performed
  1. Trans-trabecular meshwork surgery with or without an implant
  2. Trans-scleral surgery with or without implant
  3. Ciliary Body Treatment
  4. Suprachoroidal surgery with or without implant
  5. External Non Incisional Treatment

SUMMARY:
This study aims to investigate the effect of different types of glaucoma surgery on aqueous dynamics parameters (IOP, aqueous flow rate, trabecular outflow facility and uveoscleral outflow) in patients with uncontrolled open angle glaucoma or ocular hypertension (OHT)

DETAILED DESCRIPTION:
There are currently many surgical options for patients with glaucoma and ocular hypertension (OHT), including trans-trabecular meshwork surgery with or without an implant, trans-scleral surgery with or without implant, ciliary body treatment, suprachoroidal surgery with or without implant, external non-incisional treatment. However, little is known about how these different surgical techniques used to treat glaucoma affect the flow of fluid through and out of the eye (aqueous dynamics).

One hundred and fifty patients with open angle glaucoma or OHT who are deemed to require glaucoma surgery clinically will be included in a prospective interventional study to investigate the effect of a number of surgical interventions (as listed above) for glaucoma on aqueous dynamics and also to investigate the influence of baseline aqueous dynamics on the eventual outcome of the different surgical techniques. The contralateral non-operated eye will be used as control where possible.

Participants will undergo pre-operative baseline measurement of aqueous dynamics parameters (intraocular pressure (IOP), aqueous flow rate, tonographic outflow facility) 2-8 weeks after stopping to use their eye drops for glaucoma. This stopping of glaucoma drops, or treatment 'washout', is considered an intervention as it deviates from the participants' usual care. Intraocular pressure will be measured using an ocular response analyser (ORA), the outflow facility will be measured by electronic Schiøtz tonography, and the aqueous flow rate will be measured by fluorophotometry. The uveoscleral outflow will be calculated using the Goldmann equation.

Measurement of aqueous dynamics parameters will be repeated 3 months and 12 months after surgery at post-operative follow-up appointments. The follow-up measurements of aqueous dynamics parameters will also be made after 2-8 weeks treatment washout where participants have to continue to use medication for their glaucoma after the surgery. Paired student t-tests will be used to compare aqueous dynamics parameters before and after surgery.

A number of additional eye test procedures will also be performed to collect data for the study at the pre-operative baseline appointment and at routine post-operative follow-up assessments 3 months and 12 months post-surgery. Other data will be collected from eye tests that are routinely performed at the pre-operative appointment and at post-operative follow-up appointments: 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after surgery.

All the additional non-routine tests will be performed as part of standard clinical ophthalmological assessments that are routinely utilised in the ophthalmology department.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 90 (inclusive).
* Able to understand the study and give informed consent.
* Willing, able and available to participate in the study. If Flurophotometer test required must not have had prior cataract surgery.
* Diagnosis of glaucoma or OHT which requires glaucoma surgery (trans-trabecular meshwork surgery with or without an implant, trans-scleral surgery with or without implant, ciliary body treatment, suprachoroidal surgery with or without implant, external non-incisional treatment). (Defined as primary or secondary glaucoma; all types of secondary glaucoma may be included. Glaucoma will be diagnosed based on abnormal visual field testing and corresponding disc changes once seen by a glaucoma specialist.)
* It is judged clinically safe for the patient to undergo treatment washout (stop taking glaucoma drops).

Exclusion Criteria:

* Diagnostic criteria for inclusion not met.
* Allergy to fluorescein.
* It is judged as not clinically safe or patient is not willing to undergo treatment washout (stop taking glaucoma drops).
* Current use of any investigational drug or device or current participation in an interventional clinical trial/study.
* Participants in the study must be able to understand English to complete some of the tests so those who might not adequately understand written information or verbal explanations in English will not be included

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Glaucoma/OHT patients with sub-optimal intraocular pressure on multiple topical medications who require glaucoma surgical intervention to manage uncontrolled IOP.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
To investigate the effect of different types of glaucoma surgery on aqueous dynamics parameters (Intraocular Pressure IOPcc/IOPg using Ocular Response Analyzer) in patients with uncontrolled glaucoma or OHT. | 5 years
  Glaucoma surgery types (trans-trabecular meshwork surgery with or without an implant, trans-scleral surgery with or without implant, ciliary body treatment, suprachoroidal surgery with or without implant, external non-incisional treatment)
To investigate the effect of different types of glaucoma surgery on aqueous dynamics parameters (Trabecular outflow facility µL/min per mm Hg using digital schiøtz tonometer) in patients with uncontrolled glaucoma or OHT. | 5 years
  Glaucoma surgery types (trans-trabecular meshwork surgery with or without an implant, trans-scleral surgery with or without implant, ciliary body treatment, suprachoroidal surgery with or without implant, external non-incisional treatment)
To investigate the effect of different types of glaucoma surgery on aqueous dynamics parameters (Aqueous flow rate μL/min using a flurophotometer) in patients with uncontrolled glaucoma or OHT. | 5 years
  Glaucoma surgery types (trans-trabecular meshwork surgery with or without an implant, trans-scleral surgery with or without implant, ciliary body treatment, suprachoroidal surgery with or without implant, external non-incisional treatment)
To investigate the effect of different types of glaucoma surgery on aqueous dynamics parameters (Uveoscleral outflow μL/min using the Goldmann mathematical equation) in patients with uncontrolled glaucoma or OHT. | 5 years
  Glaucoma surgery types (trans-trabecular meshwork surgery with or without an implant, trans-scleral surgery with or without implant, ciliary body treatment, suprachoroidal surgery with or without implant, external non-incisional treatment)

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events | 5 years
  Glaucoma surgery types (trans-trabecular meshwork surgery with or without an implant, trans-scleral surgery with or without implant, ciliary body treatment, suprachoroidal surgery with or without implant, external non-incisional treatment)
Change in medication status from baseline | 5 years
  Glaucoma surgery types (trans-trabecular meshwork surgery with or without an implant, trans-scleral surgery with or without implant, ciliary body treatment, suprachoroidal surgery with or without implant, external non-incisional treatment)

IPD SHARING:
Plan to Share IPD: No